CLINICAL TRIAL: NCT06224348
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel Group, 3-arm, Multinational, Multicenter Study to Evaluate the Efficacy and Safety of Amlitelimab by Subcutaneous Injection in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis on Background Topical Corticosteroids
Brief Title: A Study to Evaluate the Efficacy and Safety of Subcutaneous Amlitelimab in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis on Background Topical Corticosteroids
Acronym: SHORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17561; 2023-506558-20 (Registry Identifier: CTIS); U1111-1275-9760 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Adrenal Cortex Hormones; Calcineurin Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amlitelimab dose 1 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab; Drug: Topical corticosteroids; Drug: Topical calcineurin inhibitors
- Amlitelimab dose 2 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab; Drug: Topical corticosteroids; Drug: Topical calcineurin inhibitors
- Placebo (Placebo Comparator): Subcutaneous injection as per protocol
  Interventions: Drug: Placebo; Drug: Topical corticosteroids; Drug: Topical calcineurin inhibitors

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Injection solution Route of administration: SC injection
  Other Names: SAR445229
  Arms: Amlitelimab dose 1; Amlitelimab dose 2
Drug: Placebo — Pharmaceutical form: injection solution Route of administration: SC injection
  Arms: Placebo
Drug: Topical corticosteroids — Pharmaceutical form: Topical formulation Route of administration: Topical
Drug: Topical calcineurin inhibitors — Pharmaceutical form: Topical formulation Route of administration: Topical

SUMMARY:
This is a parallel group, Phase 3, multinational, multicenter, randomized, double-blind, placebo controlled, 3-arm study for treatment of participants diagnosed with moderate-to-severe atopic dermatitis (AD) with a history of inadequate response of topical treatment, on background topical corticosteroid (TCS) and/or topical calcineurin inhibitor (TCI).

The purpose of this study is to measure the efficacy and safety of treatment with amlitelimab solution for subcutaneous (SC) injection compared with placebo in participants with moderate to severe AD aged 12 years and older on background TCS and/or TCI.

Study details include:

At the end of the treatment period, participants will have an option to enter a separate study: the blinded extension study EFC17600 (ESTUARY).

For participants not entering the blinded extension Study EFC17600 (ESTUARY), the study duration will be up to 44 weeks including a 2 to 4-week screening, a 24-week randomized double-blind period, and a 16-week safety follow-up.

For participants entering the blinded extension Study EFC17600 (ESTUARY), the study duration will be up to 28 weeks including a 2 to 4-week screening and a 24-week randomized double-blind period.

The total treatment duration will be up to 24 weeks. The total number of visits will be up to 10 visits (or 9 visits for those entering the blinded extension study EFC17600 (ESTUARY).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 12 years of age (when signing informed consent form)
* Diagnosis of AD for at least 1 year (defined by the American Academy of Dermatology Consensus Criteria)
* Documented history (within 6 months before screening) of inadequate response to topical treatments, and/or inadequate response to systemic therapies (within 12 months before screening)
* v-IGA-AD of 3 or 4 at baseline visit
* EASI score of 16 or higher at baseline
* AD involvement of 10% or more of BSA at baseline
* Weekly average of daily PP-NRS of ≥ 4 at baseline visit.
* Able and willing to comply with requested study visits and procedures
* Body weight ≥25 kg

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Skin co-morbidity that would adversely affect the ability to undertake AD assessments
* Known history of or suspected significant current immunosuppression
* Any malignancies or history of malignancies prior to baseline (with the exception of non-melanoma skin cancer excised and cured >5 years prior to baseline)
* History of solid organ or stem cell transplant
* Any active or chronic infection including helminthic infection requiring systemic treatment within 4 weeks prior to baseline
* Positive for human immunodeficiency virus (HIV), Hepatitis B or hepatitis C at screening visit
* Having active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, or who are at high risk of contracting TB
* Having received any of the specified therapy within the specified timeframe(s) prior to the baseline visit
* In the Investigator's opinion, any clinically significant laboratory results or protocol specified laboratory abnormalities at screening
* History of hypersensitivity or allergy to any of the excipients or investigational medicinal product (IMP)

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
EU, EU reference countries, and Japan: Proportion of participants with Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points at Week 24 | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
EU, EU reference countries, and Japan: Proportion of participants reaching 75% reduction from baseline in Eczema Area and Severity Index (EASI) score (EASI-75) at Week 24 | Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
US and US reference countries: Proportion of participants with vIGA-AD of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points at Week 24 | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).

SECONDARY OUTCOMES:
Proportion of participants reaching EASI-75 at Week 24 (for US and US reference countries only) | Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.
Proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) with presence of only barely perceptible erythema (no induration/papulation, no lichenification, no oozing or crusting) and a reduction from baseline of ≥2 points | Baseline to Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with ≥4-point reduction in weekly average of daily Peak Pruritus-Numerical Rating Scale (PP-NRS) from baseline in participants with baseline weekly average of daily PP-NRS ≥4 | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants reaching EASI-75 | Baseline to Week 20
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.
Proportion of participants with vIGA-AD of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points | Baseline to Week 20
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with vIGA-AD 0 (clear) | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants reaching EASI-90 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-90 is 90% reduction from baseline in EASI score.
Proportion of participants reaching EASI-100 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-100 is 100% reduction from baseline in EASI score.
Proportion of participants with PP-NRS 0 or 1 | Baseline to Week 2
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Change in Dermatology Life Quality Index (DLQI) from baseline in participants with age ≥16 years old | Baseline to Week 24
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Proportion of participants with a reduction in DLQI ≥4 from baseline in participants with age ≥16 years old and with DLQI baseline ≥4 | Baseline to Week 24
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change in Children Dermatology Life Quality Index (CDLQI) from baseline in participants with age ≥12 to <16 years old | Baseline to Week 24
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Proportion of participants with a reduction in CDLQI ≥6 from baseline in participants with age ≥12 to <16 years old and with CDLQI baseline ≥6 | Baseline to Week 24
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change in Hospital Anxiety Depression Scale (HADS) from baseline | Baseline to Week 24
  The HADS is 14-item questionnaire with two subscales: anxiety & depression. Each subscale (anxiety & depression) ranges 0-21. The total HADS score ranges 0-42 with higher score indicating a poorer state.
Proportion of participants with HADS subscale Anxiety (HADS-A) <8 in participants with baseline HADS-A ≥8 | Baseline to Week 24
  HADS-A score ranges 0-21 with higher score indicating a poorer state.
Proportion of participants with HADS subscale Depression (HADS-D) <8 in participants with HADS-D baseline ≥8 | Baseline to Week 24
  HADS-D score ranges 0-21 with higher score indicating a poorer state.
Absolute change in weekly average of daily Skin Pain-Numerical Rating Scale (SP-NRS) from baseline | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Proportion of participants with a reduction in weekly average of daily SP-NRS ≥4 from baseline in participants with baseline weekly average of daily SP-NRS ≥4 | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Absolute change in weekly average of daily Sleep Disturbance-Numerical Rating Scale (SD-NRS) from baseline | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Proportion of participants with a reduction in weekly average of daily SD-NRS ≥3 from baseline in participants with Baseline weekly average of daily SD-NRS ≥3 | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Percent change in weekly average of daily SP-NRS from baseline | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Percent change in weekly average of daily SD-NRS from baseline | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Percent change in EASI score from baseline | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Percent change in weekly average of daily PP-NRS from baseline | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Absolute change in weekly average of daily PP-NRS from baseline | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants reaching EASI-50 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score.
Proportion of participants with EASI ≤7 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Change in percent Body Surface Area (BSA) affected by AD from baseline | Baseline to Week 24
Percent change in Scoring Atopic Dermatitis (SCORAD) index from baseline | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Absolute change in SCORAD index from baseline | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Proportion of participants with a reduction in SCORAD ≥ 8.7 points from baseline in participants with baseline SCORAD score ≥ 8.7 | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Change in Patient Oriented Eczema Measure (POEM) from baseline | Baseline to Week 24
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Proportion of participants with a reduction in POEM ≥4 from baseline in participants with POEM Baseline ≥4 | Baseline to Week 24
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Proportion of participants with rescue medication use | Baseline to Week 24
Cumulative amount of topical corticosteroids (TCS) consumption | Baseline to Week 24
Percentage of TCS/topical calcineurin inhibitors (TCI) free days | Baseline to Week 24
Percentage of participants who experienced Treatment-Emergent Adverse Events (TEAEs), experienced Treatment-Emergent Serious Adverse Events (TESAEs) and/or Treatment-Emergent Adverse Events of Special Interest (AESI) | Baseline to Week 40
Serum amlitelimab concentrations | Baseline to Week 40
Incidence of antidrug antibodies (ADAs) of amlitelimab | Baseline to Week 40

CONTACTS AND LOCATIONS:
Locations (166):
- United States (40):
  - Cahaba Dermatology & Skin Health Center- Site Number : 8401066, Birmingham, Alabama
  - Johnson Dermatology- Site Number : 8401076, Fort Smith, Arkansas
  - Encino Research Center- Site Number : 8401042, Encino, California
  - Marvel Clinical Research- Site Number : 8401102, Huntington Beach, California
  - LA Universal Research Center- Site Number : 8401064, Los Angeles, California
  - Cura Clinical Research- Site Number : 8401141, Palmdale, California
  - Integrative Skin Science and Research- Site Number : 8401275, Sacramento, California
  - Southern California Dermatology- Site Number : 8401043, Santa Ana, California
  - Skin Care Research - Hollywood- Site Number : 8401071, Hollywood, Florida
  - Clever Medical Research- Site Number : 8401160, Miami, Florida
  - Acevedo Clinical Research Associates- Site Number : 8401088, Miami, Florida
  - Palm Springs Community Health Center- Site Number : 8401264, Miami Lakes, Florida
  - Global Clinical Professionals (GCP)- Site Number : 8401045, St. Petersburg, Florida
  - University of South Florida- Site Number : 8401070, Tampa, Florida
  - Avita Clinical Research- Site Number : 8401073, Tampa, Florida
  - Cleaver Medical Group- Site Number : 8401138, Dawsonville, Georgia
  - NorthShore University HealthSystem - Skokie Hospital- Site Number : 8401038, Skokie, Illinois
  - Dawes Fretzin Clinical Research- Site Number : 8401015, Indianapolis, Indiana
  - BRCR Global Gretna- Site Number : 8401243, Gretna, Louisiana
  - Velocity Clinical Research - New Orleans- Site Number : 8401155, New Orleans, Louisiana
  - Oakland Medical Center- Site Number : 8401116, Troy, Michigan
  - Allergy & Immunology Associates of Ann Arbor- Site Number : 8401078, Ypsilanti, Michigan
  - Dermatology and Skin Cancer Lee's Summit- Site Number : 8401157, Lee's Summit, Missouri
  - Skin Specialists- Site Number : 8401068, Omaha, Nebraska
  - Jubilee Clinical Research- Site Number : 8401054, Las Vegas, Nevada
  - Allcutis Research - Portsmouth- Site Number : 8401082, Portsmouth, New Hampshire
  - Equity Medical- Site Number : 8401239, New York, New York
  - Icahn School of Medicine at Mount Sinai- Site Number : 8401129, New York, New York
  - OptiSkin- Site Number : 8401163, New York, New York
  - Apex Clinical Research Center- Site Number : 8401237, Mayfield Heights, Ohio
  - Essential Medical Research- Site Number : 8401183, Tulsa, Oklahoma
  - Vial Health - DermDox Dermatology- Site Number : 8401031, Camp Hill, Pennsylvania
  - Clinical Research Center of the Carolinas- Site Number : 8401067, Charleston, South Carolina
  - SMS Clinical Research- Site Number : 8401182, Mesquite, Texas
  - Sienna Dermatology- Site Number : 8401148, Missouri City, Texas
  - Texas Dermatology and Laser Specialists- Site Number : 8401131, San Antonio, Texas
  - Discovery Clinical Trials - San Antonio - Stone Oak Parkway- Site Number : 8401026, San Antonio, Texas
  - Complete Dermatology - Sugar Land- Site Number : 8401061, Sugar Land, Texas
  - Cope Family Medicine - Ogden Clinic- Site Number : 8401114, Bountiful, Utah
  - Tanner Clinic - Layton Antelope A- Site Number : 8401151, Layton, Utah
- Argentina (10):
  - Investigational Site Number : 0320005, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320011, Buenos Aires
  - Investigational Site Number : 0320019, Buenos Aires
  - Investigational Site Number : 0320008, Buenos Aires
  - Investigational Site Number : 0320018, Buenos Aires
  - Investigational Site Number : 0320010, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320012, Corrientes
  - Investigational Site Number : 0320013, Mendoza
  - Investigational Site Number : 0320020, San Miguel de Tucumán
- Brazil (9):
  - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo- Site Number : 0760017, Vitória, Espírito Santo
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760002, Salvador, Estado de Bahia
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR- Site Number : 0760023, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760024, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto- Site Number : 0760015, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC- Site Number : 0760001, Santo André
  - Hospital Alemao Oswaldo Cruz - São Paulo- Site Number : 0760010, São Paulo
  - Hospital das Clinicas FMUSP- Site Number : 0760012, São Paulo
- Bulgaria (4):
  - Investigational Site Number : 1002007, Dupnitsa
  - Investigational Site Number : 1002004, Pleven
  - Investigational Site Number : 1002009, Sofia
  - Investigational Site Number : 1002006, Sofia
- Canada (13):
  - Investigational Site Number : 1240039, Calgary, Alberta
  - Investigational Site Number : 1240045, Red Deer, Alberta
  - Investigational Site Number : 1240046, Kamloops, British Columbia
  - Investigational Site Number : 1240030, Surrey, British Columbia
  - Investigational Site Number : 1240041, Winnipeg, Manitoba
  - Investigational Site Number : 1240057, Brampton, Ontario
  - Investigational Site Number : 1241106, Markham, Ontario
  - Investigational Site Number : 1240008, Mississauga, Ontario
  - Investigational Site Number : 1240004, Peterborough, Ontario
  - Investigational Site Number : 1240038, Richmond Hill, Ontario
  - Investigational Site Number : 1240012, Toronto, Ontario
  - Investigational Site Number : 1241107, Waterloo, Ontario
  - Investigational Site Number : 1240006, Québec, Quebec
- Chile (10):
  - Investigational Site Number : 1520009, Osorno, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520011, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520010, Santiago
  - Investigational Site Number : 1520012, Talcahuano
- China (12):
  - Investigational Site Number : 1560050, Changsha
  - Investigational Site Number : 1560060, Chengdu
  - Investigational Site Number : 1560043, Fuzhou
  - Investigational Site Number : 1560021, Guangzhou
  - Investigational Site Number : 1560044, Hangzhou
  - Investigational Site Number : 1560006, Hangzhou
  - Investigational Site Number : 1560051, Nanchang
  - Investigational Site Number : 1560005, Shanghai
  - Investigational Site Number : 1560041, Shenyang
  - Investigational Site Number : 1560047, Tianjin
  - Investigational Site Number : 1560049, Wuhan
  - Investigational Site Number : 1560003, Wuxi
- Czechia (6):
  - Investigational Site Number : 2032105, Nový Jičín
  - Investigational Site Number : 2030010, Olomouc
  - Investigational Site Number : 2032104, Ostrava
  - Investigational Site Number : 2030009, Pilsen
  - Investigational Site Number : 2030008, Prague
  - Investigational Site Number : 2030011, Prague
- France (8):
  - Investigational Site Number : 2500011, Bordeaux
  - Investigational Site Number : 2500009, Nantes
  - Investigational Site Number : 2500013, Nice
  - Investigational Site Number : 2500006, Pierre-Bénite
  - Investigational Site Number : 2500010, Romans-sur-Isère
  - Investigational Site Number : 2500012, Rouen
  - Investigational Site Number : 2500016, Saint-Pierre
  - Investigational Site Number : 2500002, Toulouse
- Germany (10):
  - Investigational Site Number : 2760020, Augsburg
  - Investigational Site Number : 2760009, Bad Bentheim
  - Investigational Site Number : 2760014, Buxtehude
  - Investigational Site Number : 2760017, Hamburg
  - Investigational Site Number : 2760021, Hamburg
  - Investigational Site Number : 2762208, Kiel
  - Investigational Site Number : 2760018, Magdeburg
  - Investigational Site Number : 2760016, Mainz
  - Investigational Site Number : 2762201, Münster
  - Investigational Site Number : 2760019, Witten
- Italy (5):
  - Investigational Site Number : 3800003, Milan, Lombardy
  - Investigational Site Number : 3800012, Bologna
  - Investigational Site Number : 3800011, L’Aquila
  - Investigational Site Number : 3800008, Pisa
  - Investigational Site Number : 3800019, Torette
- Japan (19):
  - Investigational Site Number : 3920009, Chitose, Hokkaido
  - Investigational Site Number : 3923114, Obihiro, Hokkaido
  - Investigational Site Number : 3920008, Sapporo, Hokkaido
  - Investigational Site Number : 3920006, Kobe, Hyōgo
  - Investigational Site Number : 3920005, Sagamihara, Kanagawa
  - Investigational Site Number : 3923113, Yokohama, Kanagawa
  - Investigational Site Number : 3920010, Miyagi-gun, Miyagi
  - Investigational Site Number : 3920011, Sendai, Miyagi
  - Investigational Site Number : 3923110, Sakai, Osaka
  - Investigational Site Number : 3920002, Iruma, Saitama
  - Investigational Site Number : 3923106, Mibu, Tochigi
  - Investigational Site Number : 3920004, Chūō, Tokyo
  - Investigational Site Number : 3923107, Minato, Tokyo
  - Investigational Site Number : 3920001, Tachikawa, Tokyo
  - Investigational Site Number : 3923109, Habikino
  - Investigational Site Number : 3923108, Kagoshima
  - Investigational Site Number : 3923102, Kyoto
  - Investigational Site Number : 3920003, Kyoto
  - Investigational Site Number : 3923113, Yokohama
- Spain (10):
  - Investigational Site Number : 7240019, Granada, Andalusia
  - Investigational Site Number : 7240020, Seville, Andalusia
  - Investigational Site Number : 7240008, Bilbao, Bizkaia
  - Investigational Site Number : 7240010, Esplugues de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240015, Pamplona, Navarre
  - Investigational Site Number : 7242502, Manises, Valencia
  - Investigational Site Number : 7240023, Burjassot, Valenciana, Comunidad
  - Investigational Site Number : 7242505, Alicante
  - Investigational Site Number : 7240013, Madrid
  - Investigational Site Number : 7240014, Vigo
- Turkey (Türkiye) (10):
  - Investigational Site Number : 7920010, Ankara
  - Investigational Site Number : 7920001, Antalya
  - Investigational Site Number : 7920008, Gaziantep
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920006, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920009, Istanbul
  - Investigational Site Number : 7920004, Kayseri
  - Investigational Site Number : 7920007, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17561 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25590&tenant=MT_SNY_9011